CLINICAL TRIAL: NCT03110926
Title: Induction Chemotherapy for Locally Advanced Esophageal Cancer: A Phase II Study
Brief Title: Induction Chemotherapy for Locally Advanced Esophageal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Richard Dunne, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UGIE 17037
Record Dates: First submitted 2017-03-30; First posted 2017-04-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Oxaliplatin; Leucovorin; Fluorouracil; Chemoradiotherapy; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Induction Chemotherapy /Chemoradiation (Experimental): mFOLFOX6 for 3 cycles - Oxaliplatin 85 mg/m2, 5-fluorouracil 2400mg/m2/46 hours, 5-fluorouracil bolus 400mg/m2 and leucovorin 400 mg/m2, then chemoradiation for 5 cycles - Carboplatin AUC 2mg/mL/min, Paclitaxel 50 mg/m2 and radiation therapy.
  Interventions: Drug: mFOLFOX6; Combination Product: Chemoradiation

INTERVENTIONS:
Drug: mFOLFOX6 — Induction Chemotherapy
  Other Names: Oxaliplatin; Leucovorin; 5-FU
Combination Product: Chemoradiation — Chemoradiation
  Other Names: Carboplatin; Paclitaxel; External Beam Radiation Therapy

SUMMARY:
Evaluate mFOLFOX6 (5-Fluorouracil, Leucovorin and Oxaliplatin) chemotherapy as induction treatment prior to standard neoadjuvant chemoradiation to decrease the rate of distant recurrence among patients with locally advanced esophageal cancer.

DETAILED DESCRIPTION:
The goal of the study is to evaluate mFOLFOX6 (5-Fluorouracil, Leucovorin and Oxaliplatin) chemotherapy as induction treatment prior to standard neoadjuvant chemoradiation to decrease the rate of distant recurrence among patients with locally advanced esophageal cancer. mFOLFOX6 is frequently used to treat metastatic esophageal cancer because of its high response rate in this setting. It has shown promising efficacy in several trials of patients with advanced esophageal cancer and it is the most commonly used combination regimen for this group of patients in the United States.

The investigators propose treating a sample of 40 patients with 3 cycles of induction mFOLFOX6 chemotherapy over six weeks followed by standard chemoradiation and surgery. The investigators hypothesize that patients who undergo induction chemotherapy with mFOLFOX6 prior to standard neoadjuvant chemoradiation and surgery will have a lower rate of distant disease recurrence compared to standard neoadjuvant chemoradiation and surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Must have histologically proven adenocarcinoma, squamous cell carcinoma or undifferentiated carcinoma of the esophagus, GE junction and/or gastric cardia.
2. Must have potentially resectable disease.
3. Must have ECOG performance status 0 or 1.
4. Must have adequate organ function as defined by the following criteria:

   * ANC ≥ 1,500/mm3
   * Platelet count ≥ 100,000/mm3
   * Creatinine (Cr) ≤ 1.5 mg and/or creatinine clearance ≥ 60cc/min.
   * Total bilirubin must be ≤ 1.5 x ULN unless the patient has a chronic grade 1 bilirubin elevation due to Gilbert's disease or similar syndrome due to slow conjugation of bilirubin.
   * Alkaline phosphatase must be ≤ 2 x ULN.
   * AST & ALT must be ≤ 3 x ULN.
5. Men and women of reproductive potential must agree to use an effective contraception method
6. Must be willing and able to provide written informed consent
7. Must be ≥ 18 years or older

Exclusion Criteria:

1. Prior chemotherapy, thoracic radiotherapy or prior surgical resection for an esophageal tumor.
2. Known distant metastases.
3. Patients with prior malignancies are eligible if they have been disease-free for > 5 years and are deemed by their physician to be at low risk for recurrence. Patients with squamous or basal cell carcinoma of the skin, melanoma in situ, carcinoma in situ of the cervix, or carcinoma in situ of the colon or rectum that have been effectively treated are eligible, even if these conditions were diagnosed within 5 years prior to randomization.
4. Known ≥ grade 2 neuropathy.
5. Known non-malignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude any of the study therapy drugs.
6. Known psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude them from meeting the study requirements.
7. Women who are pregnant or nursing.
8. Women and men of reproductive potential who are expecting to conceive or father children.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival rate | 2 years
  Evaluate the 2-year disease-free survival rate in patients who receive induction chemotherapy with mFOLFOX6 followed by standard chemoradiation and surgery.

SECONDARY OUTCOMES:
Pathologic examination | 2 years
  To assess, by pathologic examination of resected specimen, complete and partial response to induction chemotherapy with mFOLFOX6 followed by standard chemoradiation and surgery.
Toxicities as Assessed by CTCAE v4.0 | 25-29 weeks
  To determinate the safety and tolerability of induction chemotherapy with mFOLFOX6 followed by standard chemoradiation and surgery. Investigator will collect and record AEs as assessed by CTCAE v4.0. AEs greater than or equal to Grade 3 will be reported as means and number of participants.
Overall survival | 2 years
  Evaluate overall survival of participants who receive induction chemotherapy with mFOLFOX6 followed by standard chemoradiation and surgery.
Overall disease-free survival | 2 years
  Evaluate overall disease-free survival in patients who receive induction chemotherapy with mFOLFOX6 followed by standard chemoradiation and surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Dunne, MD, Principal Investigator — University of Rochester Wilmot Cancer Center
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Shapiro J, van Lanschot JJB, Hulshof MCCM, van Hagen P, van Berge Henegouwen MI, Wijnhoven BPL, van Laarhoven HWM, Nieuwenhuijzen GAP, Hospers GAP, Bonenkamp JJ, Cuesta MA, Blaisse RJB, Busch ORC, Ten Kate FJW, Creemers GM, Punt CJA, Plukker JTM, Verheul HMW, Bilgen EJS, van Dekken H, van der Sangen MJC, Rozema T, Biermann K, Beukema JC, Piet AHM, van Rij CM, Reinders JG, Tilanus HW, Steyerberg EW, van der Gaast A; CROSS study group. Neoadjuvant chemoradiotherapy plus surgery versus surgery alone for oesophageal or junctional cancer (CROSS): long-term results of a randomised controlled trial. Lancet Oncol. 2015 Sep;16(9):1090-1098. doi: 10.1016/S1470-2045(15)00040-6. Epub 2015 Aug 5. PMID 26254683
- [Background] Ajani JA, Komaki R, Putnam JB, Walsh G, Nesbitt J, Pisters PW, Lynch PM, Vaporciyan A, Smythe R, Lahoti S, Raijman I, Swisher S, Martin FD, Roth JA. A three-step strategy of induction chemotherapy then chemoradiation followed by surgery in patients with potentially resectable carcinoma of the esophagus or gastroesophageal junction. Cancer. 2001 Jul 15;92(2):279-86. doi: 10.1002/1097-0142(20010715)92:23.0.co;2-2. PMID 11466680
- [Background] Bains MS, Stojadinovic A, Minsky B, Rusch V, Turnbull A, Korst R, Ginsberg R, Kelsen DP, Ilson DH. A phase II trial of preoperative combined-modality therapy for localized esophageal carcinoma: initial results. J Thorac Cardiovasc Surg. 2002 Aug;124(2):270-7. doi: 10.1067/mtc.2002.122545. PMID 12167786
- [Background] Enzinger PC, Burtness BA, Niedzwiecki D, Ye X, Douglas K, Ilson DH, Villaflor VM, Cohen SJ, Mayer RJ, Venook A, Benson AB 3rd, Goldberg RM. CALGB 80403 (Alliance)/E1206: A Randomized Phase II Study of Three Chemotherapy Regimens Plus Cetuximab in Metastatic Esophageal and Gastroesophageal Junction Cancers. J Clin Oncol. 2016 Aug 10;34(23):2736-42. doi: 10.1200/JCO.2015.65.5092. Epub 2016 Jul 5. PMID 27382098
- [Background] Finley KA. Observations of bluegills fed selenium-contaminated Hexagenia nymphs collected from Belews Lake, North Carolina. Bull Environ Contam Toxicol. 1985 Dec;35(6):816-25. doi: 10.1007/BF01636593. No abstract available. PMID 4074950